CLINICAL TRIAL: NCT00823472
Title: Among IVF Patients Undergoing Fixed Antagonist Protocols With Recombinant FSH, Does Administration of Recombinant FSH From Cycle Day 5 Onwards Compared With Cycle Day 2 Onwards, Yield a Higher Number of Good Quality Embryos?
Brief Title: Trial Comparing Start Stimulation of Recombinant Follicle Stimulating Hormone (rFSH) on Cycle Day 2 Versus Cycle Day 5 in In Vitro Fertilization (IVF)
Acronym: LITE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inclusion of the study didn't go as fast as expected. Expect: 234 patients in 1 year in 2 centers. After 1,5 year only 147 patients were recruited.
Sponsor: UMC Utrecht (Other)
Collaborators: Free University Medical Center (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LITE study; CCMO: NL2370504108; METC: 08/233
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: in Vitro Fertilization; Ovulation Induction
Keywords: embryonic structures; sperm injections, intracytoplasmic; IVF; GnRH antagonist; ovarian stimulation; cycle day 2 versus cycle day 5
MeSH Terms: interventions — follitropin beta; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Start rFSH cycle day 2 (Experimental)
  Interventions: Drug: Mild stimulation
- Start rFSH on cycle day 5 (Experimental)
  Interventions: Drug: Mild stimulation

INTERVENTIONS:
Drug: Mild stimulation — Fixed daily dose of 150 IU rFSH start cycle day 5 or day 2 depending on the Arm
  Other Names: Puregon; Ganirelix

SUMMARY:
Background of the study:

Milder stimulation protocols have the advantage of being less expensive and more patient-friendly. Moreover, recent evidence suggests that mild stimulation protocols lead to lower embryo aneuploidy rates compared to conventional treatment regimens. Although with mild stimulation protocols the expected number of oocytes retrieved will be lower, pregnancy rates have shown to be similar possibly because embryo quality outfavours embryo quantity.

Objective of the study:

The aim of the study is to determine whether cycle day (CD) 5 start of stimulation will lead to better quality of embryos, based on morphology, than CD 2 start, in IVF with GnRH antagonist co-treatment started on a fixed day.

Study design:

Prospective randomized trial comparing two different starting days of ovarium stimulation (day 2 versus day 5) for IVF treatment.

Intervention:

One group wil start on cycle day 2 with stimulation of the ovaries with recombinant FSH. The other group will start on cycle day 5. Both group will start suppressing the gonadotrophin production of the the pituitary gland on cycle day 6 with a GnRH antagonist.

Primary study parameters/outcome of the study:

Primary outcome parameter is number of top embryos per ovum pick up.

Secondary study parameters/outcome of the study:

Secondary outcome measures are duration of stimulation, cancellation rate, fertilization rate, number of cumulus oocyte complexes obtained, number of mature oocytes obtained, number of top embryos per started cycle, amount of IU recFSH, and clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Female age < 36 years
* FSH < 12 IU/l
* BMI 18-29 kg/m2
* Regular cycle (25-35 days)
* No major uterine or ovarian abnormalities
* No previous IVF cycles
* Written informed consent

Exclusion Criteria:

* Oocyte donation
* Medical contra indication for pregnancy or IVF treatment
* Endometriosis ≥ grade 3
* Polycystic Ovarium Syndrome (PCOS)
* Endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney)

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart C Fauser, Prof, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- UZ Brussel, Brussels, Belgium
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Hohmann FP, Macklon NS, Fauser BC. A randomized comparison of two ovarian stimulation protocols with gonadotropin-releasing hormone (GnRH) antagonist cotreatment for in vitro fertilization commencing recombinant follicle-stimulating hormone on cycle day 2 or 5 with the standard long GnRH agonist protocol. J Clin Endocrinol Metab. 2003 Jan;88(1):166-73. doi: 10.1210/jc.2002-020788. PMID 12519847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recuited between 11-9-2008 and 1-10-2010 in both centers.
Pre-assignment Details: Patients who didn't completed the trial were cancelled before OPU due to low- or hyperresponse or before ET due to total fertilisation failure or no embryo to transfer.
Groups:
- Start rFSH Cycle Day 2: Start 150 IU rFSH subcutaneously on cycle day 2
- Start rFSH on Cycle Day 5: Start 150 IU rFSH subcutaneously on cycle day 5
Period: Overall Study
Arm/Group | Start rFSH Cycle Day 2 | Start rFSH on Cycle Day 5
Started | 80 | 67
Completed | 56 | 39
Not Completed | 24 | 28
Not completed — Physician Decision | 24 | 28

BASELINE CHARACTERISTICS:
Groups:
- Start rFSH Cycle Day 2: Start 150IU rFSH s.c. cycle day 2
- Start rFSH on Cycle Day 5: Start 150IU rFSH s.c. cycle day 5
- Total: Total of all reporting groups
Arm/Group | Start rFSH Cycle Day 2 | Start rFSH on Cycle Day 5 | Total
Number analyzed (Participants) | 80 | 67 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 67 | 147
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (3.5) | 31.1 (4.4) | 31.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 67 | 147
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 49 | 39 | 88
  Netherlands | 31 | 28 | 59

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Top Embryos Per OPU.
Description: Proportion of top embryos per ovum pick-up
Time Frame: 1 year
Population: ITT
Measure: Number; unit: percentage embryos
Arm/Group | Start rFSH Cycle Day 2 | Start rFSH on Cycle Day 5
Number analyzed (Participants) | 80 | 67
percentage embryos | 51.1 | 41.8

2. Secondary Outcome: Number of Cumulus Oocyte Complexes Obtained
Description: Number of cumulus oocyte complexes obtained after ovum pick-up
Time Frame: one year
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | Start rFSH Cycle Day 2 | Start rFSH on Cycle Day 5
Number analyzed (Participants) | 80 | 67
oocytes | 9.8 (5.4) | 8.5 (5.7)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Diary at the time of oocyte pick-up
Groups:
- Start rFSH on Cycle Day 5: Start 150IU rFSH s.c. cycle day 2=5
Arm/Group | Start rFSH Cycle Day 2 | Start rFSH on Cycle Day 5
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/67
Other Adverse Events (participants affected / at risk) | 0/80 | 0/67

LIMITATIONS AND CAVEATS:
Early termination of the trial lead to small number of subjects to be analyzed. Only half of the expected patients were included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes